CLINICAL TRIAL: NCT00552565
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Rezular (Arverapamil) in the Treatment of Irritable Bowel Syndrome With Diarrhea (IBS-D)
Brief Title: Efficacy Study of Rezular (Arverapamil) in the Treatment of Irritable Bowel Syndrome With Diarrhea (IBS-D)
Acronym: ARDIS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGI Therapeutics, Inc. (Other)
Responsible Party: David Young, AGI Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARDIS-1
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: IBS, IBS-D, R-verapamil, Arverpamil, Rezular
MeSH Terms: conditions — Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Rezular 15mg
- Rezular 37.5mg (Experimental)
  Interventions: Drug: Rezular
- Rezular - 75mg (Experimental)
  Interventions: Drug: Rezular

INTERVENTIONS:
Drug: Rezular 15mg — Oral Tablets
  Arms: 2
Drug: Placebo — placebo
  Arms: 1
Drug: Rezular — Rezular 37.5mg 3xday up to 12 weeks
  Arms: Rezular 37.5mg
Drug: Rezular — Rezular 75mg 3xday up to 12 weeks
  Arms: Rezular - 75mg

SUMMARY:
The purpose of the study is to determine the efficacy and safety of Rezular (arverapamil) in the treatment of IBS-D.

DETAILED DESCRIPTION:
We have fulfilled our enrollment requirements for this study.

This study has been designed as a multicenter, randomized, double-blind, placebo controlled parallel dose group trial. The study will be open to both women and men. At screening the patient will be assessed to see if they meet the Rome III criteria for IBS-D. After screening, patients will undergo a 14-day run-in period evaluation, during which eligibility to be randomized to drug or placebo will be determined. Patients will complete daily telephone diaries during the run-in and double-blind phases of the study. Patients will be evaluated at regularly scheduled clinic visits during double-blind phase of the study.

Patients who complete the study may have the opportunity to rollover to the open-label one-year safety study (ARDIS-3).

ELIGIBILITY:
Inclusion Criteria:

* fulfilling Rome III criteria for IBS-D

Exclusion Criteria:

* major cardiovascular disease
* psychiatric illness except mild or moderate depression
* pregnancy
* presence of other GI disease that could explain IBS-like symptoms
* history of major gastric, hepatic, pancreatic or intestinal surgery or perforation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Adequate Relief | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Wilmington, North Carolina, United States